CLINICAL TRIAL: NCT02429076
Title: Electroencephalogram Studies of Intravenous Methylphenidate-Induced Emergence From General Anesthesia
Brief Title: EEG Studies of IV Methylphenidate-Induced Emergence From Anesthesia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: We are not going to complete this study with healthy volunteers at this time.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ken Solt, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 2015P000566
Record Dates: First submitted 2015-04-08; First posted 2015-04-29 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Active Emergence From General Anesthesia
MeSH Terms: interventions — Methylphenidate; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Propofol (Experimental): Subjects in this arm will receive propofol general anesthesia
  Interventions: Drug: IV methylphenidate; Drug: Placebo; Drug: Propofol
- Sevoflurane (Experimental): Subjects in this arm will receive sevoflurane general anesthesia
  Interventions: Drug: IV methylphenidate; Drug: Placebo; Drug: Sevoflurane

INTERVENTIONS:
Drug: IV methylphenidate — IV methylphenidate will be administered to induce emergence from general anesthesia.
Drug: Placebo — normal saline
Drug: Sevoflurane — Inhaled anesthetic
  Arms: Sevoflurane
Drug: Propofol — IV anesthetic
  Arms: Propofol

SUMMARY:
The aim of this study is to test the hypothesis that methylphenidate actively induces emergence from propofol and sevoflurane general anesthesia in healthy volunteers.

DETAILED DESCRIPTION:
Basic science and clinical data suggest that activation of one or more of the brain's arousal pathways is a highly plausible way to induce active emergence from general anesthesia. The investigators have compelling experimental data demonstrating that methylphenidate is highly effective in actively inducing emergence from isoflurane and propofol general anesthesia in rodents. The available literature suggests that IV methylphenidate would be safe to administer to patients recovering from general anesthesia, and that in addition to promoting arousal, it would enhance breathing. Both of these effects would be highly desirable in patients recovering from general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-36 years
2. ASA classification 1 or 2
3. Normal body weight, BMI ≤ 30
4. Non-smoker
5. Right handed
6. No history of taking stimulants

Exclusion Criteria:

* In general, patients will be excluded from the study if the state of their chronic health problems gives them an ASA physical status classification of 3 or beyond.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Response to methlyphenidate administration | minutes to response, expected average is less than 10 minutes
  The number of minutes from the administration of methylphenidate until subjects respond to verbal commands